CLINICAL TRIAL: NCT05166967
Title: Impact of Optimal Doses of Antithymocyte Globulin Conditioning on Graft Versus-host Disease and Virus Reactivation in Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Targeted Dose Study of ATG in Haploidentical Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University People's Hospital, Peking University Institute of Hematology (Unknown); Department of Hematology, The First Affiliated Hospital of Zhengzhou University (Unknown)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2020-484-02
Record Dates: First submitted 2021-11-22; First posted 2021-12-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Haploidentical Hematopoietic Stem Cell Transplantation
Keywords: ATG; Haplo-HSCT
MeSH Terms: interventions — Antilymphocyte Serum

STUDY DESIGN:
Intervention Model Description: Random Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual dose of ATG (Experimental): Individual dose of ATG: Individual dose of ATG was Intravenous infused every day from day -5 to day -2 (total ATG dose was calculated based on pharmacokinetic index, within a range of 6 mg/kg to 13mg/kg), and the active ATG concentration ranges from 110 to 148.5UE/ml.
  Interventions: Drug: Individual Antithymocyte globulin
- Fixed dose of ATG (Active Comparator): A total amount of 10mg/kg ATG was divided into 4 days (from day -5 to day -2). The specific usage: 1.5mg/kg for day -5, 2.5mg/kg for day -4 and day -3, 3.5 mg/kg for day -2.
  Interventions: Drug: Antithymocyte globulin

INTERVENTIONS:
Drug: Individual Antithymocyte globulin — Individual dose of ATG was Intravenous infused every day from day -5 to day -2 (total ATG dose was calculated based on pharmacokinetic index, within a range of 6 mg/kg to 13mg/kg). Prophylaxis against graft versus-host disease (GVHD) was performed with cyclosporine A (CsA), mycophenolate mofetil (MMF) and short-term methotrexate.
  Arms: Individual dose of ATG
Drug: Antithymocyte globulin — A 10mg/kg total dose of antithymocyte globulin (ATG) was added to conditioning regimens for 4 days (from day -5 to day -2). Prophylaxis against graft versus-host disease (GVHD) was performed with cyclosporine A (CsA), mycophenolate mofetil (MMF) and short-term methotrexate.
  Arms: Fixed dose of ATG

SUMMARY:
The purpose of this study is to determine the response and toxicity rate of two different dosages (Individualized dosage VS. fixed dosage) of ATG as a prophylaxis for acute GVHD in haploidentical peripheral blood stem cell transplantation (haplo-PBSCT).

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGvHD) is an important complication of haploHSCT. The Seattle group initially introduced the use of ATG as a treatment for acute graft-versus-host disease (aGVHD) in allogeneic hematopoietic stem cell transplantation (haplo-PBSCT) recipients. Presently, in both myeloablative and reduced-intensity conditioning (RIC) haplo-PBSCT, ATG is part of post engraftment immunosuppressive regimens. The regimens for prophylaxis of GVHD based on 10mg/kg rabbit anti-human thymocyte immunoglobin (ATG, Thymoglobin®, Genzyme Polyclonals S.A.S) effectively reduced the occurrence of grade II-IV aGvHD. Howevre, the incidence of cytomegalovirus (CMV) and EB virus (EBV) reactivation were higher due to a slower immune reconstitution. The 100-day cumulative incidence of CMV and EBV viremia were both over 70% in our unmanipulated haplo-PBSCT program. The optimal dose of ATG balancing the efficacy of GVHD prophylaxis and the risk of virus reactivation in haplo-PBSCT remains unknown.

Reports on the pharmacokinetics of Thymoglobulin in allo-HSCT revealed a high variability. Recent pharmacokinetic studies have shown that the half-life of total ATG after transplant is longer than the active ATG (which is available to bind to human lymphocytes and causes the desired immunological effects). And active ATG appears more associated with pharmacodynamics effects. In our previous cohort study, we found that virus reactivation and acute GVHD were highly affected by ATG exposure (area under the curve, AUC). We have found an optimal range of active ATG range is 110-148.5UE/ml.day the efficacy of GVHD prophylaxis and the risk of virus reactivation. The cumulative incidence of CMV reactivation and persistent CMV hyperemia at 180 days after transplantation in the optimal total AUC group was 60.57% and 31.52% respectively. Significantly lower than 77.08% and 56.25% in the non-optimal total AUC group.

The results suggested that Individualized dosing of ATG has a potential advantage in balancing the efficacy of GVHD prophylaxis and the risk of virus reactivation in haplo-PBSCT. This may improve the survival and quality of life of patients undergoing haplo-PBSCT. A prospective randomized trial is required to compare the efficacy of Individualized dosage of ATG as a prophylaxis for acute GVHD in haplo-PBSCT.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients should have the indication of Haploidentical hematopoietic stem cell transplant.
* 2. All patients should sign an informed consent document indicating that they understand the purpose of and procedures required for the study and be willing to participate in the study.

Exclusion Criteria:

1.Patients with any conditions not suitable for the trial (investigators' decision).

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
GVHD-free and relapse-free survival (GRFS) | 12 months after transplantation
  GRFS is defined as a composite endpoint of death from any cause, disease relapse, grade III-IV acute GVHD, or moderate to severe chronic GVHD requiring systemic immunosuppression therapy.

SECONDARY OUTCOMES:
Cumulative incidences of CMV reactivation | 6 months after transplantation
  CMV reactivation was defined as DNA load ≥ 1×104 copies /mL or ≥ 1×103 copies/mL in two consecutive tests. The cumulative incidence of CMV reactivation by Day +180 post-transplantation was defined as the proportion of CMV reactivation occurring at any monitoring point during 6 months post-transplant.
Incidence of CMV disease | 6 months after transplantation
  The cumulative incidences of CMV disease in participants after transplantation,
Cumulative incidences of EBV reactivation | 6 months after transplantation
  The cumulative incidences of EBV reactivation in participants after transplantation, tested by EBV realtime PCR.
Cumulative incidences of PTLD(posttransplant lymphoproliferative disorders) | 6 months after transplantation
  The cumulative incidences of PTLD in participants after transplantation
Cumulative incidences of aGVHD | 365 days after transplantation
  The diagnosis and grading of aGVHD are based on the modified Glucksberg grading standard.
Cumulative incidences of cGVHD | 365 days after transplantation
  Chronic GVHD can be classified as "limited" or "extensive" according to the Seattle criteria, and also be classified as "mild" or "moderate" or "severe" according to the National Institutes of Health (NIH) criteria.
Neutrophil engraftment | 1 month after transplantation
  Neutrophil engraftment is defined as the first of 3 consecutive days with an absolute neutrophil count > 0.5 × 10^9/L.
Platelet engraftment | 1 month after transplantation
  Platelet engraftment is defined as the first of 7 consecutive days with an absolute platelet count > 20 × 10^9/L independent from transfusion
Overall survival (OS) | 365 days after transplantation
  Overall survival (OS) is defined as the time from randomization to death resulting from any cause.
Disease-free survival (DFS) | 365 days after transplantation
  Disease-free survival (DFS) is defined as the time from enrollment to relapse of primary disease or death from any cause, whichever occurred first.
Nonrelapse mortality (NRM) | 365 days after transplantation
  Non-relapse mortality (NRM) is defined as the time from enrollment to death of any causes other than hematologic disease relapse.
Infection rate | 365 days after transplantation
  Infection rate is defined as the proportion of participants who developed all kinds of infection

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China